CLINICAL TRIAL: NCT01453075
Title: Evaluating Three Grams Daily Valacyclovir in Patients With Chronic Hepatitis C and Herpes Simplex Virus 2 (HSV-2) Infection (Phase I)
Brief Title: Evaluating Three Grams Daily Valacyclovir in Patients With Chronic Hepatitis C and HSV-2 Infection (Phase I)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-001A-10F; 1lK2CX00536 (Other: VA CSR&D); VAL115610 (Other: VS CSR&D); NCT01525342 (obsolete NCT alias)
Record Dates: First submitted 2011-10-07; First posted 2011-10-17 (Estimated); Results first posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Hepatitis C Infection
Keywords: hepatitis C; herpes simplex type 2; veterans
MeSH Terms: conditions — Hepatitis C | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: valacyclovir (Experimental): Assigned patients will take 1.5 mg po valacyclovir twice daily
  Interventions: Drug: Valacyclovir
- Arm 2: placebo (Placebo Comparator): Assigned patients will receiving matching placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valacyclovir — Valacyclovir 1.5 mg po bid
  Arms: Arm 1: valacyclovir
Drug: Placebo — Matching placebo twice daily
  Arms: Arm 2: placebo

SUMMARY:
The purpose of this study is to study the effects of valacyclovir on patients who have hepatitis C and antibodies to herpes simplex type-2. Herpes simplex type 2 is a virus which causes genital herpes. Some persons with genital herpes have sores in their private areas but most persons do not have any symptoms at all. Valacyclovir is a medication which is commonly used to treat or prevent outbreaks of genital herpes. This medication is already approved by the Food and Drug Administration to treat genital herpes. Valacyclovir has not been approved to treat chronic hepatitis C.

The study will take 16 weeks. Participants will be assigned to take either the study drug, valacyclovir, or a sugar pill that looks exactly like valacyclovir. The researchers and the persons participating will not know which medication they are receiving. Study visits will occur every two weeks and will take approximately 3-45 minutes. All study visits will occur at the G.V. Sonny Montgomery VA Medical Center.

DETAILED DESCRIPTION:
Study is a randomized, double-blinded, placebo-controlled, Phase II clinical trial. Participants will be recruited while attending regularly scheduled clinic appointments at the Jackson VA Medical Center. Baseline Visit. Participants will be randomized 1:1 in groups of 10 to receive valacyclovir 1.5 gram orally twice daily or matching placebo. Enrolled participants will complete 12 weeks of assigned therapy.

At the initial visit, participants will complete a short questionnaire detailing past medical/social history and relevant symptoms. Venipuncture will be performed to obtain samples for the laboratory tests. The baseline de-identified serum sample will be obtained from the clinical lab and stored in research-approved freezer space for future confirmation with the Biokit HSV-2 rapid assay. Follow-up visits will be scheduled at two-week intervals after baseline. At each visit, pill-count, compliance and tolerability of medications will be assessed using a short questionnaire. Venipuncture will be performed every four weeks (i.e., at every other follow-up visit) to provide samples for the tests described below. Information from each study visit will be recorded into the chart by the PI or Research Assistant (RA) and entered into an encrypted database on a VA server. Laboratory Tests. HSV-2 infection will be confirmed by performing the Biokit HSV-2 rapid assay on the baseline stored serum sample using methods previously described in this proposal. Laboratory tests will include 1) complete blood count, comprehensive metabolic profile, and quantitative hepatitis C virus (HCV) RNA; and 2) Focus HerpeSelect HSV-1 Immunoglobulin G (IgG) for participants who were seronegative for HSV-1 at baseline. Patient's IL28-B genotype will also be assessed at baseline. The PI will review all laboratory parameters.

Baseline characteristics between the groups will be compared using appropriate parametric tests. Analysis will be intention to treat with the inclusion of all subjects who were randomized to drug or placebo. The primary outcome is change in HCV viral load in the treatment group compared with placebo. Because the investigators are expecting a 0.5 log10 decline in HCV viral load, the investigators will use one-sided parametric tests. All viral loads will be log10-transformed before analysis.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of chronic HCV infection with genotype testing and previous positive HerpeSelect HSV-2 IgG assay

Exclusion Criteria:

* Antiherpes or immunomodulatory therapy during the past 30 days
* HIV or chronic hepatitis B infection
* Decompensated liver disease (ascites, hepatic encephalopathy, coagulopathy, jaundice/icterus)
* Creatinine clearance < 50 ml/min.
* Female subject who is pregnant or nursing
* Gastrointestinal disorder which might result in malabsorption of valacyclovir
* History of erythema multiforme major, thrombotic thrombocytopenia purpura or hemolytic uremic syndrome
* Therapy for hepatitis C in the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-11; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Burton, MD, Principal Investigator — G.V. (Sonny) Montgomery VA Medical Center, Jackson, MS
Locations (1):
- G.V. (Sonny) Montgomery VA Medical Center, Jackson, MS, Jackson, Mississippi, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Valacyclovir | Arm 2: Placebo
Started | 16 | 15
Completed | 11 | 14
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Valacyclovir | Arm 2: Placebo | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (3.5) | 58.8 (3.5) | 58.8 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Effect of HSV-2 Suppression on HCV Viral Load.
Description: Measure the change in serum HCV viral load at baseline and 12 weeks in patients who have chronic hepatitis C and HSV-2 infection who receive the 3 grams daily valacyclovir versus placebo
Time Frame: baseline; 12 weeks
Population: Analyzed patients who completed study
Measure: Mean (Standard Error); unit: log(IU/mL)
Arm/Group | Arm 1: Valacyclovir | Arm 2: Placebo
Number analyzed (Participants) | 11 | 14
log(IU/mL) | .18 (.104) | .03 (.75)

ADVERSE EVENTS:
Arm/Group | Arm 1: Valacyclovir | Arm 2: Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No